CLINICAL TRIAL: NCT05045859
Title: A Multimethod Psych-physiological Randomized Controlled Trial of a Couples' Intervention for PTSD
Brief Title: A Couples' Intervention Protocol for PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Prof. Rachel Dekel, prof., Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11022021
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Psychological Trauma
Keywords: post traumatic stress disorder; Cognitive-Behavioral Conjoint Therapy (CBCT); couples therapy; cognitive behavioral therapy (CBT); heart rate variability (HRV); Randomized controlled trial; telepsychology; conference video
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The study will be based on an RCT design. The screening process will consist of an initial phone call and two video conference sessions, to assess eligibility. Eligible Couples will be randomized using block randomization for assignment to two conditions: A CBCT and a waitlist (WL) control. The WL group will be assigned to CBCT after the waiting period. The design includes four points of assessment: Pre-treatment/pre-WL (baseline) (T1); during treatment/waiting period (T2 - different measures at various intervals); post-treatment/post-waiting period (T3); and at a 4-month follow-up (T4). Self- report measures will be administered at all time-points. A dyadic communication lab interaction will be conducted at T1 & T3. At T2, PTSD and marital satisfaction will be measured in every session. physiological monitoring will be conducted at T1 and T3, and at six out of 15 sessions. qualitative interviews with a randomly selected sub-sample (N=12) will take place at T1 and T3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, therapists, investigators and outcome assesors are blind to the condition the individual participant was assigned to, by encrypting the names of the individual into a number-letter codes.The therapists led the intervention group was not aware of the participants condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBCT for PTSD (Experimental): CBCT for PTSD is a 15-session, manualized therapy developed by Monson and Fredman, designed to simultaneously improve PTSD symptoms and enhance relationship functioning.
  Interventions: Behavioral: CBCT for PTSD
- No Intervention: Wait- List Controls (WL) (No Intervention): Patients in wait- list control arm received no active treatment during their 15-weeks waiting period. At the end of that period received the exact intervention as the study group.

INTERVENTIONS:
Behavioral: CBCT for PTSD — CBCT for PTSD is a 15-session, manualized therapy developed by Monson and Fredman, designed to simultaneously improve PTSD symptoms and enhance relationship functioning. It assumes that PTSD exists within the couple's relationship and that partners can join together to reduce the presence of PTSD in their relationship. Sessions are organized into three phases of treatment: (1) psychoeducation about PTSD and relationships; (2) behavioral interventions to enhance relationship functioning; and (3) dyadic cognitive intervention designed to contextualize trauma memories and address trauma-relevant cognitions held by either partner that keep the PTSD and/or relationship distress alive. Out-of-session assignments are designed to assist the couple in reinforcing skills learned in the sessions.
  Arms: CBCT for PTSD

SUMMARY:
Posttraumatic stress disorder (PTSD) is a multifaceted disorder resulting from intense and/or life-threatening trauma. PTSD sequelae often have a ripple effect on close others, including spouses and children. Studies report high levels of relationship distress for both those with PTSD and their partners as well as emotional distress. Despite the extensive knowledge on the effects of PTSD on couple relations and vice versa, and the limitations of individual therapies in addressing these issues, there has been a major lag in the development and study of couples' interventions in the context of PTSD. the current study will examine the efficacy of Cognitive Behavioral Conjoint Therapy (CBCT) for PTSD. It will employ an RCT to examine both outcomes and processes of change via multiple methods of assessment, including self-report questionnaires, qualitative interviews and physiological co-regulation measures. Moreover, it will employ a modified procedure via video conference due to COVID-19 in addition to in-person treatment option. The study will therefore contribute to theoretical understandings of the effects of PTSD on couples, to the development of therapies specifically intended for such couples.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a multifaceted disorder resulting from intense and/or life-threatening trauma. PTSD sequelae often have a ripple effect on close others, including spouses and children. Despite the extensive knowledge on the effects of PTSD on couple relations and vice versa, and the limitations of individual therapies in addressing these issues, there has been a major lag in the development and study of couples' interventions in the context of PTSD.

The current study will examine the efficacy of Cognitive Behavioral Conjoint Therapy (CBCT) for PTSD. It will employ RCT design to examine both outcomes and processes of change via multiple methods of assessment, including self-report questionnaires, qualitative interviews, and physiological co-regulation measures. Moreover, it will employ a modified procedure via video conference due to COVID-19.

The first aim is to examine the efficacy of CBCT using multiple methods in RCT design in the Israeli context. The following hypotheses related to treatment efficacy will be examined:

1. The investigators expect that the CBCT group will show a larger decrease in the level of patient PTSS and a decrease in depression, anxiety, anger, guilt and marital aggression among both partners in comparison to the waiting list (WL) controls. Marital satisfaction of both partners is expected to increase.
2. The investigators expect that each of the spouses will gradually, over the course of treatment, show more regulated autonomic nervous system (ANS) activity (e.g., GSR, HRV, RSA) among the CBCT group; The investigators also expect more positive physiological co-regulation between spouses over time.

2. The second aim of the study is to understand change processes and mechanisms specific to CBCT. The following hypotheses will be examined:

1. The investigators will examine the mediating role of accommodation, emotional regulation, self-disclosure and partner responsiveness: compared to WL controls, CBCT will be associated with higher levels of these factors in mid-treatment, and they in turn will be associated with better outcomes (e.g., PTSS, depression, marital adjustment) post-treatment.
2. The investigators expect that synchrony levels between the couples will rise after CBCT. In addition, (2.a) The investigators expect PTSD severity and marital satisfaction to moderate these associations: Among couples where the individual with PTSD has more severe PTSD and where couples report on lower levels of marital satisfaction, the change in the level of arousal and strength of physiological synchrony will be lower.
3. The investigators expect that synchrony levels between the couples will rise from session to session. The investigators will also explore the dynamics of change in physiological co-regulation during sessions, as they correspond with different components of the intervention protocol. In addition The investigators will explore the association between synchronicity to the study's main outcomes (e.g., PTSS, depression, marital adjustment) post-treatment.

(3.b) The investigators will examine the role of accommodation as a mediator of change in the level of physiological co-regulation before and after the intervention. Thus, compared to WL controls, those in CBCT will show more accommodation over time, which in turn will be associated with higher levels of synchrony/co-regulation.

As for the qualitative design, it does not assume hypotheses, but rather poses questions. A sub-sample of 15 couples will undergo a semi-structured qualitative interview regarding their subjective experience in therapy, before and after the intervention. The interview will consist of pre-defined open-ended questions regarding 4 main elements: 1. The expectations and the experience of couples' therapy via video conference. 2. Assessing the impact and effectiveness of the intervention on couples relationship and psychological distress; 3. Changes that occurred in spouses' mutual understanding of PTSD, its effects on the relationship, and how they handle and react in light of these effects. This will give participants a chance to describe their experiences over the course of therapy in their own words. In this part of the study, there is one directional hypothesis: The investigators expect interviews to reflect a positive experience from therapy, reflecting both symptomatic change (in PTSS) and positive changes in couples' adjustment and relationship.

The study is a randomized controlled trial (RCT), including 60 couples (120 participants in total) in which one of the spouses suffers from PTSD. An initial phone prescreen will be conducted to determine possible eligibility for all potential participants who respond or are referred via various recruitment strategies. The phone prescreen will be used to provide initial information about the study and the assessment procedures, as well as initial Screening method to assess level of motivation and relationship status. Individuals who appear eligible will then be contacted for two longer screening sessions with a trained staff member, via video conference, to further assess eligibility based on the exclusion criteria. During the screening sessions, participants will be sent an electronic consent form. Participants will be asked to complete an online survey collecting demographic information, self-report questionnaires and the Clinicians Administered PTSD Scale for DSM-V. The self report questionnaires will assess: (a) active psychosis; (b) substance use; (c) suicidal risk; (d) physical, verbal or cyber aggression in the relationship. Participants data will be collected through Qualtrics, an online data-capture tool. Participants excluded for significant suicidal ideation, psychosis or substance abuse will be referred to appropriate treatment options. Couples found to be eligible will receive a thorough explanation about the treatment, the study and its various components, and will subsequently be randomized using a block randomization method for assignment.

The couples will be randomly assigned to 2 conditions: (1) Group CBCT (n=30), (2) Waitlist control group, subsequently assigned to treatment (n=30). The CBCT intervention will be conducted remotely through video conference. As the study continues, participants may be given the option to choose between remote therapy and face-to-face meetings, depending on the state of COVID-19 spread in Israel. Participants will complete structured clinical interview and self-report questionnaires tapping psychological (PTSD symptoms, depression, anger), behavioral (domestic violence), and marital satisfaction; As well as physiological measures (HRV and skin conductance) at 4 assessments: pre-/during/post- treatment, and 4 months after treatment.

To date, no RCT has examined CBCT for PTSD in Israel or examined the treatments efficacy when sessions take place in a telehealth platform. In addition, The study will be the first study to examine physiological co-regulation changes due to CBCT for PTSD. Therefore, the study will contribute to theoretical understandings of the effects of PTSD on couples, to the development of therapies specifically intended for such couples. and finally, to the well-being of Israeli PTSD patients and their spouses.

ELIGIBILITY:
Inclusion Criteria:

1. have a cohabiting partner or spouse and both spouses must commit to staying in the relationship through 15 sessions of CBCT for PTSD
2. have a current diagnosis of PTSD based on Diagnostic and Statistical Manual of Mental Disorders (5th Edition [DSM-5]; [2]), assessed with the Clinician Administered PTSD Scale for DSM-5 (CAPS-5;80)
3. not participate in concurrent psychotherapies directly targeting PTSD (e.g., eye movement desensitization and reprocessing; present centered therapy; PE) or concurrent couples therapy

Exclusion Criteria:

1. unmanaged active psychosis or manic episode (assessed with Yale University PRIME Screening Test)
2. substance use disorder warranting primary substance use treatment or detoxification (assessed with AUDIT;109 and DAST-10;110])
3. Imminent suicidal risk (assessed with Paykel questionnaire;111)
4. severe physical, verbal or cyber aggression currently or in the past 3 months (assessed with CARS;112 and CTS-2;84)
5. a current PTSD diagnosis for both spouses (assessed with CAPS-5;80).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS-5) | 8 months
  The CAPS-5 (80) is a structured clinical interview designed to assess PTSD. A life-event checklist of traumatic events included in the instrument allows for an assessment of trauma history. Each question on the CAPS-5 corresponds to a DSM-5 criterion for PTSD. Diagnosis used the severity score cutoff of 2 (moderate/threshold) or greater on a scale ranging from 0 (absent) to 4 (extreme). The number of symptoms that meet the cutoff within each subscale is then compared against diagnostic criteria to determine whether a PTSD diagnosis is appropriate. Moreover, the CAPS-5 includes items assessing social, occupational, and overall impairment, global PTSD symptom severity, and validity of the individual report.
PTSD Checklist (PCL-5) | 8 months
  The PCL-5 is a 20-item self-report questionnaire assessing PTSD symptom severity based on DSM-V criteria. Items are rated on a five-point scale ranging from 0 (not at all) to 4 (extremely). The PCL-5 is well validated, with good internal consistency, test-retest reliability, and convergent and discriminant validity
Physiological couples' co-regulation | 4 months
  Physiological monitoring of both partners will be conducted at T1 and T3, as well as in 6 therapy sessions. Physiological measures will be assessed using the MindWare Mobile Recorder, that is aimed at monitoring autonomic balance, cardiac performance, respiratory measurements, and respiratory activity. Both spouses are fitted with specialized electrodes to measure ECG (for the derivation of HRV), and GSR (for the derivation of electrodermal activity from the skin).
  At T1, to assess a baseline level of physiological co-regulation the study will utilize a lab-based method with stationary physiological equipment. Participants will complete an adapted videotaped dyadic interaction before and after the intervention. Couples will share and discuss a negative context: the effects of the PTSD on their relationship; and a positive context: a positive experience they've undergone together.
Dyadic Adjustment Scale (DAS) | 8 months
  A 32-item measure of relationship quality. The scale is divided into 4 subscales:
  1. Dyadic Consensus - degree to which respondent agrees with partner
  2. Dyadic Satisfaction -- degree to which respondent feels satisfied with partner
  3. Dyadic Cohesion -degree to which respondent and partner participate in activities together
  4. Affectional Expression -degree to which respondent agrees with partner regarding emotional affection. higher scores represent greater relationship satisfaction.

SECONDARY OUTCOMES:
The Patient Health Questionnaire-9 (PHQ-9) | 8 months
  PHQ-9 is a self-administered questionnaire used to assess major depression symptoms, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It can yield either a continuous score, or a probable major depressive disorder diagnosis using a cut-off of 10. The sensitivity and specificity of the PHQ-9 compare favorably with structured psychiatric interviews and the Cronbach alpha was found to be 0.89 in a sample of primary care patients.
Difficulties in Emotion Regulation (DERS) | 8 months
  Self-report questionnaire designed to test difficulties in the emotional regulation process. The questionnaire contains 36 items that relate to awareness of emotions and emotional reactions
Perceived Partner Responsiveness (PPR) | 8 months
  Self-report questionnaire used to assess people's perception of their partners responsiveness. Participants rated items on a 9-point Likert scale (1 = not at all true, 9 = completely true). Items with higher scores indicating greater perceived partner responsiveness.
the self-disclosure index (SDI) | 8 months
  Self-disclosure assesses the extent of disclosure in 10 topic areas. Participants completed the scale items on a 6-point Likert scale (1= discuss not at all, 6= discuss fully and completely) in regard to how much they disclosed to the partner.
Conflict Tactic Scale (CTS) | 8 months
  The CTS-2 measures psychological and physical attacks on a partner in a dating, cohabiting, or marital relationship and also the use of negotiation or reasoning to deal with conflicts. The CTS-2 is a 42-item scale, containing 5 subscales (negotiation, psychological aggression, physical assault, sexual coercion and physical injury) and is usually administered to both partners. The scale requires respondents to report the number of times they committed specific behavior in the past year and how many times their partner had committed the same behavior (Straus 2004). For the purpose of our research we only interviewed women and used victimization items for psychometric analyses.
  The items are rated on an 8-point frequency scale ranging from never to more than 20 times (Straus et al. 1996). The CTS-2 provides rates of ever prevalence and annual incidence of spousal violence, as well as chronicity and severity for the aspects of spousal conflict.
Brief Symptom Inventory (BSI) | 8 months
  The BSI-18 items were designed to measure three dimensions of psychiatric disorders: somatization (SOM), depression (DEP), and anxiety (ANX). Each of the three subscales was measured by six items, respectively. All BSI-18 items used a 5-point, Likert-type response option format (0 - not at all; 1 - a little bit; 2 - moderately; 3 -quite a bit; 4 - extremely)
the State-Trait Anger Expression Inventory (STAXI) | 8 months
  The STAXI provides a self-reported measure of the experience and expression of anger in 44 items. Individuals answered on a 4-point Likert scale (score range: 0-132) to assess either the intensity of their angry feelings or the frequency in which anger is experienced, expressed, or controlled
Post Traumatic Growth Inventory (PTGI) | 8 months
  the self-report questionnaire is used to measure the positive psychological changes that resulted from experiencing a traumatic event. Participants are asked to indicate the degree to which a positive change had occurred in their life as a result of their experience. Each statement used a 6-point Likert-type scale from not at all (0) to a very great degree (5), with a potential range of scores from 0-105. The PTGI consists of 21 statements with five discrete factors: relating to others, spiritual or religious changes, a renewed appreciation of life, personal strength, and new possibilities.
Trauma Related Guilt Inventory (TRGI) | 8 months
  The self-report questionnaire is a 32-item self-report measure that assesses the cognitive and emotional aspects of guilt associated with a traumatic event. The TRGI generates three scales-Global Guilt, Distress, and Guilt Cognitions-and three subscales (Hindsight Bias, Wrongdoing, and Lack of Justification); with response options ranging from 0 (not at all true) to 4 (extremely true).
post traumatic cognition inventory (PTCI-9) | 8 months
  The PTCI-9 is a 9-item self-report measure that asks participants to rate their agreement or disagreement with statements about their thoughts and beliefs related to a traumatic event. Participants rate the degree to which they agree or disagree with each statement using a 7-point scale ranging from 1 (totally disagree) to 7 (totally agree).
Significant Others Response to Trauma (SORTS) | 8 months
  The SORTS is a self-report measure designed to assess partner behaviors performed in relation to the identified patient's PTSD symptoms. Items on the SORTS consist of two parts: First, partners are asked to rate the frequency with which they engaged in each behavior within the past month on a scale from 0 (never) to 4 (daily or almost every day). Second, partners are asked to rate either the extent to which engaging in the behavior distressed them on a scale from 0 (not at all) to 4 (extremely) or the amount of effort they exerted engaging in each behavior on a scale from 0 (none) to 4 (extremely high amount). Four items (i.e., 3, 4, 11, 18) include a "not applicable" option, which is recoded as 0 before the items are totaled. Items are summed to yield a total score, frequency subscale score, and intensity subscale score.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Dekel, Prof., Principal Investigator — Bar Ilan University
Locations (1):
- Bar- Ilan University, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
IPD would be available to other researchers, including Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report and Analytic Code through e- mail or publications.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Kulka RA, Schlenger WE, Fairbank JA, Hough RL, Jordan BK, Marmar CR, et al. Trauma and the Vietnam War Generation: Report of Findings from the National Vietnam Veterans Readjustment Study. New York: Brunner/Mazel; 1988.
- [Background] Skodol AE, Schwartz S, Dohrenwend BP, Levav I, Shrout PE, Reiff M. PTSD symptoms and comorbid mental disorders in Israeli war veterans. Br J Psychiatry. 1996 Dec;169(6):717-25. doi: 10.1192/bjp.169.6.717. PMID 8968629
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Thorp SR, Stein MB. Post-traumatic stress disorder and functioning. PTSD Res Q. 2005;16(3):1- 8.
- [Background] Lambert JE, Engh R, Hasbun A, Holzer J. Impact of posttraumatic stress disorder on the relationship quality and psychological distress of intimate partners: a meta-analytic review. J Fam Psychol. 2012 Oct;26(5):729-37. doi: 10.1037/a0029341. Epub 2012 Aug 27. PMID 22924422
- [Background] Taft CT, Watkins LE, Stafford J, Street AE, Monson CM. Posttraumatic stress disorder and intimate relationship problems: a meta-analysis. J Consult Clin Psychol. 2011 Feb;79(1):22-33. doi: 10.1037/a0022196. PMID 21261431
- [Background] Miller MW, Wolf EJ, Reardon AF, Harrington KM, Ryabchenko K, Castillo D, Freund R, Heyman RE. PTSD and conflict behavior between veterans and their intimate partners. J Anxiety Disord. 2013 Mar;27(2):240-51. doi: 10.1016/j.janxdis.2013.02.005. Epub 2013 Mar 4. PMID 23523947
- [Background] Riggs DS, Byrne CA, Weathers FW, Litz BT. The quality of the intimate relationships of male Vietnam veterans: problems associated with posttraumatic stress disorder. J Trauma Stress. 1998 Jan;11(1):87-101. doi: 10.1023/A:1024409200155. PMID 9479678
- [Background] LaMotte AD, Taft CT, Reardon AF, Miller MW. Agreement between veteran and partner reports of intimate partner aggression. Psychol Assess. 2014 Dec;26(4):1369-74. doi: 10.1037/pas0000018. Epub 2014 Sep 29. PMID 25265413
- [Background] Lunney CA, Schnurr PP. Domains of quality of life and symptoms in male veterans treated for posttraumatic stress disorder. J Trauma Stress. 2007 Dec;20(6):955-64. doi: 10.1002/jts.20269. PMID 18157892
- [Background] Monson CM, Fredman SJ. Cognitive-Behavioral Conjoint Therapy: Harnessing the Healing Power of Relationships. New York, NY: Guilford Press; 2012.
- [Background] Glynn SM, Eth S, Randolph ET, Foy DW, Urbaitis M, Boxer L, Paz GG, Leong GB, Firman G, Salk JD, Katzman JW, Crothers J. A test of behavioral family therapy to augment exposure for combat-related posttraumatic stress disorder. J Consult Clin Psychol. 1999 Apr;67(2):243-51. doi: 10.1037//0022-006x.67.2.243. PMID 10224735
- [Background] Monson CM, Macdonald A, Fredman SJ, Schumm JA, Taft C. Empirically supported couple and family therapies for PTSD. In: Friedman MJ, Terence MK, editors. Handbook of PTSD: Science and Practice, 2nd ed. New York, NY: The Guilford Press; 2014. p. 451-65.
- [Background] Trautmann S, Wittchen HU. Trauma and PTSD in Europe. In: Marmar CB, Nemeroff CR, editors. Post-Traumatic Stress Disorder. New York, NY: Oxford University Press; 2018. p. 133-46.
- [Background] Sexton T, Gordon KC, Gurman A, Lebow J, Holtzworth-Munroe A, Johnson S. Guidelines for classifying evidence-based treatments in couple and family therapy. Fam Process. 2011 Sep;50(3):377-92. doi: 10.1111/j.1545-5300.2011.01363.x. PMID 21884076
- [Background] Rodgers B, Elliott R. Qualitative methods in psychotherapy outcome research. In: Gelo O, Pritz A, Rieken B, editors. Psychotherapy Research: Foundations, Process, and Outcome. Vienna: Springer-Verlag; 2015. p. 559-78.